CLINICAL TRIAL: NCT06207877
Title: An Investigation of the Effect of Cagrilintide and Semaglutide Combination Treatment(CagriSema) on Energy Intake, Appetite and Gastric Emptying in People With Overweight or Obesity
Brief Title: A Research Study to Look at How CagriSema Influences Food Intake, Appetite and Emptying of the Stomach in People With Excess Body Weight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9838-4695; U1111-1286-0585 (Other: World Health Organization (WHO)); 2023-504792-24-00 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — cagrilintide; semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CagriSema (Experimental): Participants will receive dose 1 cagrilintide and dose 2 semaglutide subcutaneously once-weekly (dose escalation period of 16 weeks) during the maintenance period of 5 weeks.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide
- Placebo (Active Comparator): Participants will receive placebo matched to cagrilintide and semaglutide subcutaneously once-weekly for 21 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cagrilintide — Cagrilintide will be administered subcutaneously.
  Arms: CagriSema
Drug: Semaglutide — Semaglutide will be administered subcutaneously.
  Arms: CagriSema
Drug: Placebo — Placebo will be administered subcutaneously.
  Arms: Placebo

SUMMARY:
This research study tests if CagriSema influences food intake, appetite and emptying of the stomach in people with excess body weight. Participant will either get CagriSema (active medicine) or placebo (a dummy medicine), which has no effect on the body. The treatment participants get is decided by chance. The study will last for about 32 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Aged 18-65 years (both inclusive) at the time of signing informed consent.
* Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.
* Body mass index (BMI) equal to or above 27.0 kilograms per meter square (kg/m^2) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator.

Exclusion Criteria:

* Glycated haemoglobin (HbA1C) greater than or equal to (≥) 6.5 % (48 millimoles per mole [mmol/mol]) at screening.
* History of type 1 or type 2 diabetes mellitus.
* Any clinically significant body weight change (≥5% self-reported change) or dieting attempts (e.g., participation in a weight reduction program) within 90 days before screening.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using highly effective contraceptive method.
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, gastrointestinal, or endocrinological conditions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Relative change in energy intake during ad libitum lunch, evening meal and snackbox | Baseline to Day 156
  Measured in percentage (%).

SECONDARY OUTCOMES:
Change in energy intake during ad libitum lunch, evening meal and snackbox | Baseline to Day 156
  Measured in kilojoule (KJ).
Change in amount of food consumed during ad libitum lunch, evening meal and snackbox | Baseline to Day 156
  Measured in grams (g).
AUC0-5h,para, area under the paracetamol concentration-time curve from 0 to 5 hours after start of standardised meal | Day 1 and Day 155: 0-5 hour after standardised meal
  Measured in hour*milligram per milliliter ( h*mg/mL).
AUC0-1h,para, area under the paracetamol concentration-time curve from 0 to 1 hour after start of standardised meal | Day 1 and Day 155: 0-1 hour after standardised meal
  Measured in h*mg/mL.
Cmax,para, maximum observed paracetamol concentration | Day 1 and Day 155: 0-5 hour after standardised meal
  Measured in microgram per milliliter (µcg/mL).
tmax,para, time to maximum observed paracetamol concentration after start of standardised meal | Day 1 and Day 155: 0-5 hour after standardised meal
  Measured in hours (h).
Change in percent energy intake of high fat, sweet food in total ad libitum energy intake in the evening snack box | Baseline to Day 156
  Measured in %-point.
Change in Control of Eating questionnaire (COEQ): Craving Control score | Baseline to Day 154
  The Control of Eating Questionnaire (COEQ) is a self-reported measure assessing various aspects of eating behaviour and related psychological factors. The COEQ has 19 different questions designed to assess the intensity and type of food cravings, as well as subjective sensations of appetite and mood. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control (0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); Higher score represents a greater level of Craving Control.
Change in COEQ: Positive Mood score | Baseline to Day 154
  The COEQ is a self-reported measure assessing various aspects of eating behaviour and related psychological factors. The COEQ has 19 different questions designed to assess the intensity and type of food cravings, as well as subjective sensations of appetite and mood. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control (0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); Higher score represents a greater level of Craving Control.
Change in COEQ: Craving for Sweets score | Baseline to Day 154
  The COEQ is a self-reported measure assessing various aspects of eating behaviour and related psychological factors. The COEQ has 19 different questions designed to assess the intensity and type of food cravings, as well as subjective sensations of appetite and mood. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control (0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); Higher score represents a greater level of Craving Control.
Change in COEQ: Craving for Savoury food score | Baseline to Day 154
  The COEQ is a self-reported measure assessing various aspects of eating behaviour and related psychological factors. The COEQ has 19 different questions designed to assess the intensity and type of food cravings, as well as subjective sensations of appetite and mood. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control (0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); Higher score represents a greater level of Craving Control.
Change in mean postprandial Visual Analogue Scale (VAS) ratings of Hunger | Baseline to Day 156
  Measured in millimeter (mm). VAS appetite questions record the participants' sensations within Hunger, Satiety, Fullness, Prospective food consumption by the participants on a paper printed scale line from 0 to 100 mm. The appetite score will be calculated as [hunger + (100 - satiety) + (100 - fullness) + prospective food consumption]/4. Scores of 0 mm are worst and scores of 100 mm are best.
Change in mean postprandial VAS ratings of Fullness | Baseline to Day 156
  Measured in mm. VAS appetite questions record the participants' sensations within Hunger, Satiety, Fullness and Prospective food consumption by the participants on a paper printed scale line from 0 to 100 mm. The appetite score will be calculated as [hunger + (100 - satiety) + (100 - fullness) + prospective food consumption]/4. Scores of 0 mm are worst and scores of 100 mm are best.
Change in mean postprandial VAS ratings of Satiety | Baseline to Day 156
  Measured in mm. VAS appetite questions record the participants' sensations within Hunger, Satiety, Fullness and Prospective food consumption by the participants on a paper printed scale line from 0 to 100 mm. The appetite score will be calculated as [hunger + (100 - satiety) + (100 - fullness) + prospective food consumption]/4. Scores of 0 mm are worst and scores of 100 mm are best.
Change in mean postprandial VAS ratings of Prospective food consumption | Baseline to Day 156
  Measured in mm. VAS appetite questions record the participants' sensations within Hunger, Satiety, Fullness and Prospective food consumption by the participants on a paper printed scale line from 0 to 100 mm. The appetite score will be calculated as [hunger + (100 - satiety) + (100 - fullness) + prospective food consumption]/4. Scores of 0 mm are worst and scores of 100 mm are best.
Change in mean postprandial VAS ratings of Appetite Score | Baseline to Day 156
  Measured in mm. VAS appetite questions record the participants' sensations within Hunger, Satiety, Fullness and Prospective food consumption by the participants on a paper printed scale line from 0 to 100 mm. The appetite score will be calculated as [hunger + (100 - satiety) + (100 - fullness) + prospective food consumption]/4. Scores of 0 mm are worst and scores of 100 mm are best.
Change in Power of Food questionnaire for Food available score | Baseline to Day 155
  The Power of Food questionnaire measures three factors that correspond to different levels of food proximity and reflect responsiveness to food-abundant environments: food available (food that is available, but not physically present), food present (food that is present, but not tasted), and food tasted (food that is tasted, but not consumed). Moreover, an aggregate score is calculated as the mean of the three subdomains. The questionnaire consists of 15 questions, and the participants will be asked to rate their agreement or disagreement with each statement on a 5-point scale (ranging from "strongly disagree" to "strongly agree").
Change in Power of Food questionnaire for Food present score | Baseline to Day 155
  The Power of Food questionnaire measures three factors that correspond to different levels of food proximity and reflect responsiveness to food-abundant environments: food available (food that is available, but not physically present), food present (food that is present, but not tasted), and food tasted (food that is tasted, but not consumed). Moreover, an aggregate score is calculated as the mean of the three subdomains. The questionnaire consists of 15 questions, and the participants will be asked to rate their agreement or disagreement with each statement on a 5-point scale (ranging from "strongly disagree" to "strongly agree").
Change in Power of Food questionnaire for Food tasted score | Baseline to Day 155
  The Power of Food questionnaire measures three factors that correspond to different levels of food proximity and reflect responsiveness to food-abundant environments: food available (food that is available, but not physically present), food present (food that is present, but not tasted), and food tasted (food that is tasted, but not consumed). Moreover, an aggregate score is calculated as the mean of the three subdomains. The questionnaire consists of 15 questions, and the participants will be asked to rate their agreement or disagreement with each statement on a 5-point scale (ranging from "strongly disagree" to "strongly agree").
Change in Power of Food questionnaire for Composite score | Baseline to Day 155
  The Power of Food questionnaire measures three factors that correspond to different levels of food proximity and reflect responsiveness to food-abundant environments: food available (food that is available, but not physically present), food present (food that is present, but not tasted), and food tasted (food that is tasted, but not consumed). Moreover, an aggregate score is calculated as the mean of the three subdomains. The questionnaire consists of 15 questions, and the participants will be asked to rate their agreement or disagreement with each statement on a 5-point scale (ranging from "strongly disagree" to "strongly agree").
Change in mean score from the Monetary Choice Questionnaire | Baseline to Day 157
  The 27-item version of the Monetary Choice Questionnaire63 is used to assess participants' individual preference for immediate versus delayed monetary rewards. The questions comprise hypothetical choices between smaller immediate rewards or larger delayed rewards. The specific amounts and delays of the rewards vary across questions. For each question, the participant is asked to choose which option they would prefer. The responses are used to calculate a measure of participants' willingness to delay gratification and their discount rate (k) for delayed rewards.
Change in body weight | Baseline to Day 155
  Measured in %.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S'
Locations (1):
- Parexel International GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com